CLINICAL TRIAL: NCT04425213
Title: Obesity as a Risk Factor for Mortality of Critically Ill Patients With Coronavirus Disease 2019 (COVID-19): a Cohort Study of the First Wave in Nancy, France
Brief Title: Obesity and Mortality of Critically Ill Patients With COVID-19
Acronym: COV-OB-ICU
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI082
Record Dates: First submitted 2020-05-28; First posted 2020-06-11 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-05

CONDITIONS: COVID; Severe Acute Respiratory Syndrome; Obesity; Comorbidities and Coexisting Conditions
Keywords: Mortality; Covid-19; Invasive mechanical ventilation; Obesity; Acute Respiratory Distress syndrome; Intensive Care Unit; Critically ill patient
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Obesity; COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal weight: BMI < 25 kg/m2
- Overweight: BMI : 25 - 29.9 kg/m2
- Moderate obesity: BMI : 30 - 39.9 kg/m2
- Severe obesity: BMI : > or = 40 kg/m2

SUMMARY:
Disproportionate impact of COVID-19 in patients with obesity is now well established.

Obesity is associated with severe forms of COVID-19 and may be a risk factor of intensive care unit (ICU) admission. Obesity is associated with COVID-19 related hospital death in a large United Kingdom cohort study. However, there is a gap of knowledge on assessment of outcomes such as severity of Acute Respiratory Distress syndrome (ARDS), duration of hospitalisation and mortality in ICU. Moreover, an obesity survival paradox has been observed in patients with ARDS. This raises the question whether the obesity paradox has been broken by COVID-19.

The investigators aim to explore risk factors of in-ICU death for patient with COVID-19, including obesity and other chronic diseases and to describe the clinical course and outcomes, including the management of acute respiratory failure and other intensive care management.

DETAILED DESCRIPTION:
The investigators aim to report ICU mortality for patients according to BMI category and to describe the detailed ICU clinical course of illness :

* Risk factors for ICU mortality : age, sex, baseline comorbidities
* Causes of death
* Risk factors for use of non invasive mechanical ventilation
* Non-fatal outcomes
* Ventilator-free days
* ICU length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with COVID-19 pneumonia admitted to ICUs between February 27th and April 18th 2020.
* Infection confirmed by reverse transcriptase polymerase chain reaction assay or radiologically by chest computed tomography scan

Exclusion Criteria:

* No weight or height measurement available in the medical files

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to ICUs of the University Hospital during the first Covid -19 wave in Nancy, Région Grand Est, France
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
ICU mortality | through study completion, an average of 14 days
  number of fatal cases

SECONDARY OUTCOMES:
Invasive mechanical ventilation | through study completion, an average of 14 days
  number of patients with invasive mechanical ventilation
In-hospital mortality | through study completion, an average of 21 days
  number of fatal cases

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Ziegler, PU-PH, Principal Investigator — CHRU of Nancy
Locations (1):
- Centre hospitalo-universitaire régional de Nancy, Vandœuvre-lès-Nancy, France